# Study of APRV and ICP in Patients with Severe Traumatic Brain Injury

NCT 02507973

Date: 3/24/15

## Introduction

Management of patients with Traumatic Brain Injury (TBI) emphasizes on prevention of secondary insults such as hypotension and hypoxemia which negatively impact outcomes <sup>1</sup>. Both hypotension <sup>2-4</sup> and hypoxemia <sup>5,6</sup> are not only independent risk factors for increased mortality in patients with TBI, but also lead to increased intracranial pressure (ICP), which is also another independent risk factor for high mortality <sup>4,7-10</sup>.

All patients with severe TBI (Glasgow Coma Scale ≤8) require sedation and mechanical ventilation for airway protection, oxygenation and minimization of obnoxious stimuli which may elevate ICP <sup>11</sup>. Mechanical ventilation, however, carries risks of increasing intrathoracic pressure, airway pressure (Paw) and may lead to increased ICP <sup>12,13</sup>.

Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that switches between high ( $P_{High}$ ) and low ( $P_{Low}$ ) continuous positive airway pressure while allowing spontaneous breathing at both phases. Alveolar recruitment and oxygenation occur during  $P_{High}$  whereas ventilation occurs during brief releases to  $P_{Low}^{14,15}$ . APRV has been used successfully in patients with multisystem trauma <sup>16-19</sup>. However literature about APRV and patients with severe TBI has been scant as concern that APRV with high positive airway pressure could result in elevated ICP still exists.

Dart et al  $^{16}$  showed that APRV could be used to improve oxygenation among multisystem trauma patients with ARDS or acute lung injuries, without affecting airway pressure (Paw). The authors informally mentioned that several patients with TBI in their studies tolerated APRV well without increasing ICP. Nemer et al reported that pressure-controlled recruitment maneuver with peak pressure up to  $50 \text{ cm H}_2\text{O}$  for 2 minutes did not increase ICP in patients with subarachnoid hemorrhage  $^{20}$ . A single case report published successful oxygenation of a hypoxemic patient with subarachnoid hemorrhage using APRV without increase of patient's ICP  $^{21}$ . In addition to improving oxygenation, APRV was also shown to improve cerebral blood flow and spinal blood flow in animals undergoing APRV with spontaneous breathing  $^{22}$ .

## **Hypothesis**

Therefore, we hypothesize that APRV could be safely used in patients with severe TBI as it does not increase their ICP and compromising their Cerebral Perfusion Pressure (CPP), while preventing hypoxemia and hypercapnia in these patients.

# **Project Primary Goal**

This pilot study, to the best of our knowledge, is the first study that specifically investigates the efficacy of APRV among patients with severe TBI. We aim to investigate whether APRV can safely oxygenate patients without compromising their ICP and CPP.

## **Study Personnel**

Principal Investigator: Dr. Debora Stein

Co-investigator: Ms. Claire Rosen (point of contact)

Drs. Thomas Grissom, Quincy Tran, Molly Deane, Michael Anstadt, Peter Hu, Darren Zimmerman, Sara Murthi, Maureen McCunn, Dadjati Bajadia.

## Study Methodology

#### Methods:

We will conduct an observational crossover study. We aim to recruit 50 patients with severe TBI requiring intracranial pressure monitoring during their stay at the Neuro Trauma ICU at the R Adams Cowley Shock Trauma Center. Each patient at admission will initially receive a primary mode of mechanical ventilation as determined by the attending trauma intensivists.

12-18 hours after recruitment, continuous monitoring of patients' ICP and hemodynamic status (ICP, HR, RR, SpO<sub>2</sub>, EtCO<sub>2</sub>, MAP, CPP, SpO<sub>2</sub>, and EtCO<sub>2</sub>) will commence to collect patients' baseline data for 30 minutes. Patients will then undergo low tidal volume mechanical ventilation (LOTV), serving as a control mode of ventilation, for 2 hours prior to switching back to the primary mode of ventilation for 30 minutes. Next, patients will be placed on APRV for 2 hours. While receiving APRV, patients' ICP and hemodynamic status will be continuously monitored and recorded for comparison and analysis. After 2 hours of APRV, patients will be switched back to their previous mode of ventilation and more data are collected for another 30 minutes. This sequence of ventilation is illustrated in figure 1.

Intracranial pressure will be measured every 15 minutes during the study period. While undergoing low tidal volume ventilation and APRV, patient's volume statuses and cardiac functions will also be assessed using a non-invasive, non-radioactive modality such as Transthoracic Echocardiography.

Figure 1. Sequence of mechanical ventilation and data collection.



Figure 2. Flow chart of APRV Protocol:



Figure 3. Flow Chart for LOTV protocol



#### Inclusion Criteria

- Intracranial pressure monitoring
- Mechanically ventilated

#### **Exclusion Criteria**

- Age < 18</li>
- Pregnant women
- Prisoners
- Initial mode of ventilation = APRV
- Providers' judgments

#### Consent:

The patients will not be able to consent for themselves, due the severity of their conditions. We will seek consent from legally authorized representative if available or patients' next-of-kin.

#### Outcomes

- Primary outcome: ICP
- Secondary outcomes: MAP, CPP, SpO2, EtCO<sub>2</sub>, any interventions for ICP or for hemodynamic instability.

# **Analysis Plan**

### Data Security:

Patient's data will be recorded on a standardized Microsoft Excel spreadsheet. This spreadsheet will first be password-protected, then encrypted by commercial 128-bit encryption software (<a href="www.boxcryptor.com">www.boxcryptor.com</a>). The encrypted spreadsheet then will be stored in a secure, password-protected online storage with extra security designed for corporation (OneDrive for Business by Microsoft Corporation, Redmond WA; <a href="https://onedrive.live.com/about/en-nz/business/">https://onedrive.live.com/about/en-nz/business/</a>).

These measures of security allow maximal collaborations between investigators while enhancing safety for patients' protected health information.

# Data Analysis:

We aim to report our findings as following:

| Table 1. Patient Demographics |
|----------------------------------------|
| Number of patients |
| Age (years) |
| Gender |
| BMI |
| Mechanism of injury |
| Motor vehicle collision, n (%) |
| Gunshot wound, n (%) |
| Fall, n (%) |
| GCS score |
| ISS |
| Primary mode of mechanical ventilation |
| PaO2/FiO2 ratio |
| ICU length of stay (days) |
| Hospital length of stay (days) |
| Mortality |

| Table 2. Outcome Measurements | | | | | | |
|---|---|---|---|---|---|---|
| Dependent Measure<br>(Mean, Interquartile) | Baseline | LOTV | APRV | Conventional MV | | <i>p</i> -value |
| | | | | Pre-<br>APRV | Post-<br>APRV | |
| ICP | | | | | | |
| MAP | | | | | | |
| CPP | | | | | | |
| CVP | | | | | | |
| Heart Rate | | | | | | |
| Respiratory Rate | | | | | | |
| SpO <sub>P</sub> | | | | | | |
| EtCO <sub>2</sub> | | | | | | |
| Volume status by TTE | | | | | | |
| Therapeutic | | | | | | |
| interventions for ICP, | | | | | | |
| blood pressure | | | | | | |

| Table 3. Adverse Events |
|-------------------------|
| Patients not |
| tolerating APRV |
| N, (%) |

| Causes | Elevated ICP |
|--------|--------------|
| N, (%) | CPP < 50 |
| | Hypoxemia |
| | Hypercapnia |
| | Tachycardia |

All continuous variables will be reported as mean with interquartile values (IQR).

# **Estimated Study Length**

There were 1259 patients with isolated blunt TBI (Abbreviated Injury Scale of brain was  $\geq$  2 while AIS for other body region was  $\leq$  2) admitted to the R Adams Cowley Shock Trauma Center in 2013. Therefore, we estimate that we will be able to recruit 2-3 patients per week.

Our pilot study is expected to finish recruitment within 6-8 months.

# **Target Conferences**

The American Association for the Surgery of Trauma: Sept. 09-12, 2015

The Society of Critical Care Medicine 44<sup>th</sup> Congress: January 17-21, 2015

# Budget:

None

#### References

- 1. Brain Trauma Foundation, American Association of Neurological Surgeons, Congress of Neurological Surgeons, et al. Guidelines for the management of severe traumatic brain injury. I. blood pressure and oxygenation. *J Neurotrauma*. 2007;24 Suppl 1:S7-13. doi: 10.1089/neu.2007.9995 [doi].
- 2. Chesnut RM, Marshall SB, Piek J, Blunt BA, Klauber MR, Marshall LF. Early and late systemic hypotension as a frequent and fundamental source of cerebral ischemia following severe brain injury in the traumatic coma data bank. *Acta Neurochir Suppl (Wien)*. 1993;59:121-125.
- 3. Fearnside MR, Cook RJ, McDougall P, McNeil RJ. The westmead head injury project outcome in severe head injury. A comparative analysis of pre-hospital, clinical and CT variables. *Br J Neurosurg*. 1993;7(3):267-279.
- 4. Schreiber MA, Aoki N, Scott BG, Beck JR. Determinants of mortality in patients with severe blunt head injury. *Arch Surg.* 2002;137(3):285-290. doi: soa1149 [pii].
- 5. Jones PA, Andrews PJ, Midgley S, et al. Measuring the burden of secondary insults in head-injured patients during intensive care. *J Neurosurg Anesthesiol*. 1994;6(1):4-14.
- 6. Stocchetti N, Furlan A, Volta F. Hypoxemia and arterial hypotension at the accident scene in head injury. *J Trauma*. 1996;40(5):764-767.
- 7. Brain Trauma Foundation, American Association of Neurological Surgeons, Congress of Neurological Surgeons, et al. Guidelines for the management of severe traumatic brain injury. VIII. intracranial pressure thresholds. *J Neurotrauma*. 2007;24 Suppl 1:S55-8. doi: 10.1089/neu.2007.9988 [doi].

- 8. Marshall LF, Smith RW, Shapiro HM. The outcome with aggressive treatment in severe head injuries. part I: The significance of intracranial pressure monitoring. *J Neurosurg*. 1979;50(1):20-25. doi: 10.3171/jns.1979.50.1.0020 [doi].
- 9. Saul TG, Ducker TB. Effect of intracranial pressure monitoring and aggressive treatment on mortality in severe head injury. *J Neurosurg*. 1982;56(4):498-503. doi: 10.3171/jns.1982.56.4.0498 [doi].
- 10. Narayan RK, Kishore PR, Becker DP, et al. Intracranial pressure: To monitor or not to monitor? A review of our experience with severe head injury. *J Neurosurg*. 1982;56(5):650-659. doi: 10.3171/jns.1982.56.5.0650 [doi].
- 11. Brain Trauma Foundation, American Association of Neurological Surgeons, Congress of Neurological Surgeons, et al. Guidelines for the management of severe traumatic brain injury. XI. anesthetics, analgesics, and sedatives. *J Neurotrauma*. 2007;24 Suppl 1:S71-6. doi: 10.1089/neu.2007.9985 [doi].
- 12. Nyquist P, Stevens RD, Mirski MA. Neurologic injury and mechanical ventilation. *Neurocrit Care*. 2008;9(3):400-408. doi: 10.1007/s12028-008-9130-7 [doi].
- 13. Stevens RD, Lazaridis C, Chalela JA. The role of mechanical ventilation in acute brain injury. *Neurol Clin*. 2008;26(2):543-63, x. doi: 10.1016/j.ncl.2008.03.014 [doi].
- 14. Daoud EG. Airway pressure release ventilation. *Annals of Thoracic Medicine*. 2007;2(4):176-179. doi:10.4103/1817-1737.36556.
- 15. Dart BW,4th, Maxwell RA, Richart CM, et al. Preliminary experience with airway pressure release ventilation in a trauma/surgical intensive care unit. *J Trauma*. 2005;59(1):71-76. doi: 00005373-200507000-00010 [pii].

- 16. Maung AA, Luckianow G, Kaplan LJ. Lessons learned from airway pressure release ventilation. *J Trauma Acute Care Surg.* 2012;72(3):624-628. doi: 10.1097/TA.0b013e318247668f [doi].
- 17. Maxwell RA, Green JM, Waldrop J, et al. A randomized prospective trial of airway pressure release ventilation and low tidal volume ventilation in adult trauma patients with acute respiratory failure. *J Trauma*. 2010;69(3):501-10; discussion 511. doi: 10.1097/TA.0b013e3181e75961 [doi].
- 18. Andrews PL, Shiber JR, Jaruga-Killeen E, et al. Early application of airway pressure release ventilation may reduce mortality in high-risk trauma patients: A systematic review of observational trauma ARDS literature. *J Trauma Acute Care Surg.* 2013;75(4):635-641. doi: 10.1097/TA.0b013e31829d3504 [doi].
- 19. Nemer SN, Caldeira JB, Azeredo LM, et al. Alveolar recruitment maneuver in patients with subarachnoid hemorrhage and acute respiratory distress syndrome: A comparison of 2 approaches. *J Crit Care*. 2011;26(1):22-27. doi: 10.1016/j.jcrc.2010.04.015 [doi].
- 20. Marik PE, Young A, Sibole S, Levitov A. The effect of APRV ventilation on ICP and cerebral hemodynamics. *Neurocrit Care*. 2012;17(2):219-223. doi: 10.1007/s12028-012-9739-4 [doi].
- 21. Kreyer S, Putensen C, Berg A, et al. Effects of spontaneous breathing during airway pressure release ventilation on cerebral and spinal cord perfusion in experimental acute lung injury. *J Neurosurg Anesthesiol*. 2010;22(4):323-329. doi: 10.1097/ANA.0b013e3181e775f1 [doi].

Daoud EG. Airway pressure release ventilation. *Annals of Thoracic Medicine*. 2007;2(4):176-179. doi:10.4103/1817-1737.36556.